CLINICAL TRIAL: NCT02335229
Title: A Post Market Observational Cohort Study to Assess the Performance of the Spinal Modulation Dorsal Root Ganglion Stimulator System for the Management of Chronic Post Surgical Pain
Brief Title: A Post Market Study to Assess the Spinal Modulation Dorsal Root Ganglion Stimulator System in Chronic Post Surgical Pain
Status: Terminated | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-SMI-2013
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-01

CONDITIONS: Chronic Post Surgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Axium DRG Neurostimulator: All eligible subjects recruited and treated with the Axium Neurostimulator
  Interventions: Device: Axium DRG Neurostimulator

INTERVENTIONS:
Device: Axium DRG Neurostimulator — Implantation with Axium DRG Neurostimulator

SUMMARY:
20-SMI-2013 is a post market, observational, questionnaire based study to assess the effectiveness of the commercially available Axium neurostimulator in the management of chronic post surgical pain

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Chronic post surgical pain for at least 6 months
4. Failed conservative treatments for chronic pain including but not limited to pharmacological therapy, physical therapy and interventional pain procedures for chronic pain
5. Minimum baseline pain rating of 60 mm on the Visual Analog Scale in the primary region of pain
6. Subject is able to provide written informed consent
7. Pain medication dosage has been stable for at least 30 days
8. Patient has been included for implantation according to standard criteria from the Dutch Neuromodulation Society

Exclusion Criteria:

1. Female subject of childbearing potential is pregnant/nursing, plans to become pregnant or is unwilling to use approved birth control
2. Escalating or changing pain condition within the past month as evidenced by investigator examination
3. Subject has had corticosteroid therapy at an intended site of stimulation within the past 30 days
4. Subject has had radiofrequency treatment of an intended target Dorsal Root Ganglion within the past 3 months
5. Subject currently has an active implantable device including implantable cardioverter defibrillator, pacemaker, spinal cord stimulator or intrathecal drug pump
6. Subject is unable to operate the device
7. Subjects with indwelling devices that may pose an increased risk of infection
8. Subjects currently has an active infection
9. Subject has participated in another clinical investigation within 30 days
10. Subject has a coagulation disorder or uses anticoagulants that, in the opinion of the investigator, precludes participation
11. Subject has been diagnosed with cancer in the past 2 years.
12. Patient has no other exclusion criteria according to standard criteria from the Dutch Neuromodulation Society

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient suffering from chronic post surgical pain
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Academisch Medisch Centrum, Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Subjects: All subjects enrolled into the study with intent to treat with the Axium Neurostimulator
Period: Overall Study
Arm/Group | All Enrolled Subjects
Started | 30
Received Trial System | 10
Received Permanent System | 26
Completed | 23
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 50 [18 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity for Overall Pain From Pre-treatment Baseline
Description: The Visual Analog Scale (VAS) is self-administered instrument assessing average pain intensity. Subjects rated their pain on a horizontal line, 10 cm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher pain level. The values range from 0 (minimum pain) to 10 (maximum pain).
Time Frame: Baseline, 3, 6, 12 and 24-Month Visits
Population: Differences in participants over time is due to early withdrawals and missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Subjects Treated With the Permanent Implantable Axium System: All subjects treated with the Axium implantable neurostimulator
Arm/Group | Subjects Treated With the Permanent Implantable Axium System
Number analyzed (Participants) | 30
units on a scale
  Baseline: number analyzed (Participants) | 28
  Baseline | 6.7 (2.0)
  3-Month Visit: number analyzed (Participants) | 25
  3-Month Visit | 5.2 (2.5)
  6-Month Visit: number analyzed (Participants) | 18
  6-Month Visit | 3.9 (2.7)
  12-Month Visit: number analyzed (Participants) | 20
  12-Month Visit | 4.8 (2.6)
  24-Month Visit: number analyzed (Participants) | 21
  24-Month Visit | 4.8 (2.0)

2. Primary Outcome: Percentage of Subjects With at Least 50% Pain Reduction
Description: Percent of subjects with at least a 50% reduction. The Visual Analog Scale (VAS) is self-administered instrument assessing average pain intensity. Subjects rated their pain on a horizontal line, 10 cm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher pain level. The values range from 0 (minimum) to 10 (maximum).
Time Frame: 3, 6, 12 and 24-Month Visits
Population: Differences in participants over time is due to early withdrawals and missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With the Permanent Implantable Axium System
Number analyzed (Participants) | 30
Participants
  3-Month Visit: number analyzed (Participants) | 25
  3-Month Visit | 6
  6-Month Visit: number analyzed (Participants) | 18
  6-Month Visit | 5
  12-Month Visit: number analyzed (Participants) | 20
  12-Month Visit | 5
  24-Month Visit: number analyzed (Participants) | 21
  24-Month Visit | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Informed Consent through study exit (24-Month visit).
Arm/Group | All Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 8/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=30)
Increasing pain due to lead failure/malfunction (Product Issues) | 1 (1)
Low blood sodium level (Investigations) | 1 (1)
Lead damaged due to accidental incision (Injury, poisoning and procedural complications) | 1 (1)
Malignant tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=30)
Broken lead (Product Issues) | 1 (1)
IPG migration (Product Issues) | 1 (1)
Lead migration (Product Issues) | 2 (2)
Pain at IPG Pocket (General disorders) | 3 (3)
Partial loss of stimulation and pain at IPG pocket (Product Issues) | 1 (1) — These Adverse Events were monitored/assessed in such a manner that the specific Adverse Event Terms cannot be separated.
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bleeding/Hematoma (Vascular disorders) | 4 (4)
Dura Puncture (Injury, poisoning and procedural complications) | 1 (1)
Foot injury (Injury, poisoning and procedural complications) | 1 (1)
Increased pain in the target area (General disorders) | 1 (1)
Kicking movement during the night (Nervous system disorders) | 1 (1)
Loss of stimulation (Product Issues) | 2 (2)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Tap (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-05-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT02335229/Prot_SAP_000.pdf